CLINICAL TRIAL: NCT00215839
Title: A Multi-Center, Randomized, Open-Label, Phase IIIb Study Investigating the Safety and Efficacy of Peginterferon a-2a Plus Ribavirin for the Treatment of Chronic Hepatitis C Infection in HIV Infected Persons Who Have Failed to Achieve a Sustained Virologic Response Following Previous Interferon Therapy
Brief Title: HRN 004- Peginterferon a-2a Plus Ribavirin for Chronic Hepatitis C Infection in HIV Infected Persons Who Have Failed to Achieve a Sustained Virologic Response Following Previous Interferon Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hepatitis Resource Network (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRN 004
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis C Infection in HIV Infected Persons; HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Ribavirin

INTERVENTIONS:
Drug: Peginterferon a-2a plus Ribavirin

SUMMARY:
Objectives:

Primary To evaluate the safety, tolerability, and efficacy of Peginterferon a-2a plus Ribavirin for the treatment of chronic hepatitis C (CHC) infection in persons co-infected with human immunodeficiency virus (HIV) who have failed to achieve a sustained virologic response following previous interferon therapy.

Secondary

* To evaluate the virological response to Peginterferon a-2a plus Ribavirin at weeks 12 and 24 as compared to baseline values.
* To evaluate the sustained virological response Peginterferon a-2a plus Ribavirin at post-treatment weeks 4, 12, and 24 as compared to baseline.
* To evaluate the histological effects of long-term Peginterferon a-2a therapy through comparison of liver biopsy results following 96 weeks of Peginterferon a-2a therapy to baseline values.
* To evaluate the safety and tolerability of long-term Peginterferon a-2a therapy in patients who have previously failed to achieve a sustained virologic response following interferon therapy.
* To investigate the effects of long-term Peginterferon a-2a therapy on clinical outcomes of HIV disease.

Study Design:

All qualifying patients will enter the treatment phase and be dosed as follows:

Peginterferon a-2a 180mg by subcutaneous route once weekly plus

Ribavirin:

* 800 mg (400 mg bid) if body weight < 65 kg
* 1000 mg (400 mg a.m. and 600 mg p.m.) if body weight > 65 kg and < 85 kg
* 1200 mg (600 mg bid) if body weight > 85 kg

Patients with undetectable levels of HCV-RNA at Treatment Week 24 will continue on previously assigned Peginterferon a-2a plus Ribavirin combo-therapy for an additional 24 weeks. Patients with detectable levels of HCV-RNA will be randomized to Peginterferon a-2a mono-therapy or no treatment for 72 weeks.

* Group A: Peginterferon a-2a 90mg mono-therapy for 72 weeks.
* Group B: No CHC therapy for 72 weeks

All patients entering the study are required to have a baseline liver biopsy (within 18 months of study entry). Patients entering the 72-week randomized arm of the trial will have a post-study liver biopsy upon completion of the trial.

Study Population:

100 HIV infected adults with chronic hepatitis C infection who have failed to achieve a sustained virologic response following previous interferon therapy.

Dosage and Administration:

Combo-therapy: Peginterferon a-2a 180mg by subcutaneous route once weekly plus

Ribavirin:

* 800 mg (400 mg bid) if body weight < 65 kg
* 1000 mg (400 mg a.m. and 600 mg p.m.) if body weight > 65 kg and < 85 kg
* 1200 mg (600 mg bid) if body weight > 85 kg Mono-therapy: Peginterferon a-2a 90mg in 1mL solution administered subcutaneously once weekly.

Efficacy Evaluations:

Laboratory analysis, liver biopsies, quality of life assessments, and changes in Peginterferona-2a and Ribavirin dosages will be obtained.

Safety Evaluations:

* Assessment of laboratory evaluations
* vital signs
* incidence and severity of adverse experiences
* dose adjustments
* premature withdrawal for safety reasons
* progression of disease as measured by HCV viral load
* AIDS defining events

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this trial, patients must have documentation of the following:

4.2.1 Written informed consent specific to this protocol obtained prior to screening and willingness to participate in and comply with the study.

4.2.2 Male and female patients >18 years of age.

4.2.3 Detectable plasma HCV-RNA by RT-PCR or other assay (bDNA).

4.2.4 HCV genotype result must be available at screening (historical determinations of genotype are acceptable).

4.2.5 Evidence of HIV infection (reactive HIV antibody with Western blot confirmation).

4.2.6 Chronic liver disease consistent with chronic hepatitis C infection on a biopsy, as judged by a qualified pathologist, obtained within the past 18 months. For all participants, both the liver biopsy report and the biopsy specimen (both an H and E slide and a Trichrome slide) must be made available for review by the central pathologist.

4.2.7 Previous antiviral treatment with alfa interferon monotherapy or, or interferon alfa plus ribavirin combination therapy administered for at least 12 weeks with the failure to obtain a sustained virologic response.

4.2.8 No therapy with interferon or interferon plus ribavirin or other specific anti-HCV medications within 4 weeks of the screening.

4.2.9 Compensated liver disease with the following laboratory parameters at screening (results within 1 month of screening):

* Hemoglobin values of ³ 11 gm/dL
* WBC ³ 3,000/mm3
* Neutrophil count ³1,250/mm3
* Platelets ³ 70,000/mm3
* Prothrombin time £ 3 seconds prolonged compared to control, or equivalent INR ratio
* Bilirubin within 20% of the upper limit of normal (unless non-hepatitis related factors such as Gilbert's disease or the use of indinivir explains an indirect bilirubin rise).
* Albumin ³ 3.0 g/dL
* Serum creatinine £ 1.4 mg/dL
* Fasting blood sugar £ 115 mg/dL for non-diabetic patients
* Hemoglobin A1C £ 8.5% for diabetic patients (whether on medication and/or diet controlled)

4.2.10 Thyroid Stimulating Hormone (TSH) within normal limits or thyroid disease under clinical control (within 3 months of screening)

4.2.11 Alpha-fetoprotein (AFP) value within normal limits obtained within the prior year. For patients with results above the upper limit of normal but < 100 ng/mL both of the following are required:

* Alpha-fetoprotein value < 100 ng/mL obtained within 3 months prior to entry AND
* Ultrasound obtained within 3 months prior to entry that is negative for evidence of hepatocellular carcinoma.

4.2.12 CD4 T cell count and HIV RNA level (by RT-PCR) within 4 weeks of screening:

* CD4 <100 Eligible with HIV RNA <25,000 by RT-PCR
* CD4 > 100 - Eligible with any HIV RNA level by RT-PCR

4.2.13 Stable antiretroviral regimen of FDA-approved agents for at least 4 weeks prior to baseline or has taken no antiretroviral agents within 4 weeks prior to baseline.

4.2.14 Reconfirmation and documentation that all sexually active female patients of childbearing potential are practicing adequate contraception (intrauterine device, oral contraceptives, progesterone implanted rods [Norplant], medroxyprogesterone acetate [Depo-Provera], surgical sterilization, barrier method [diaphragm + spermicide], or monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide) during the treatment period and for 6 months after discontinuation of therapy. Female patients must not breast feed during the treatment period and for 6 months after discontinuation of therapy. A urine pregnancy test obtained at entry prior to the initiation of treatment must be negative.

4.2.15 Reconfirmation and documentation that sexually active male patients are practicing acceptable methods of contraception (vasectomy, use of a condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 6 months after discontinuation of therapy.

4.2.16 Anyone at high risk of coronary artery disease should have a stress test performed prior to entry. This would include, but not be limited to, patients over age 55 who have a history of ischemia or who have a significant history of hypertension, diabetes mellitus, obesity, smoking and/or strong family history of coronary artery disease. Patients with evidence of ischemia on resting or stress EKG, or a history of an arrhythmia, angina or a myocardial infarction within 12 months must be excluded.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for this trial:

4.3.1 Inability or unwillingness to provide written informed consent specific to this protocol or unwillingness to participate in and comply with the study.

4.3.2 Women with ongoing pregnancy or breast feeding.

4.3.3 Male partners of women who are pregnant.

4.3.4 Hypersensitivity to interferon or ribavirin.

4.3.5 Evidence of advanced liver disease such as a history of or presence of ascites, bleeding varices, or spontaneous encephalopathy.

4.3.6 Any other causes for chronic liver disease other than chronic hepatitis C.

4.3.7 Hemoglobinopathies (e.g., Thalassemia) or any other cause of hemolytic anemia.

4.3.8 Any known preexisting medical condition that could interfere with the patient's participation in the protocol including: CNS trauma or active seizure disorders requiring medication; poorly controlled diabetes mellitus; serious pulmonary disease; immunologically-mediated diseases; gout; or any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.

4.3.9 Patients with evidence of ischemia on stress testing (required for patients at risk of or with a history of coronary artery disease, ECG evidence of ischemia, an arrhythmia, cardiac failure, coronary surgery, uncontrolled hypertension, angina or a myocardial infarction within 12 months.

4.3.10 Active or acute HIV-related opportunistic infection.

4.3.11 Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration)

4.3.12 History of major organ transplantation with an existing functional graft (including Bone Marrow Transplants)

4.3.13 History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) £6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.

4.3.14 Concomitant medication with, rifampin/rifampicin, rifabutin, pyrazinamide, isoniazid, ganciclovir, thalidomide, oxymetholone (Anadrolâ), and immunomodulatory treatments (including supraphysiologic doses of steroids).

4.3.15 Evidence of alcohol and/or drug abuse within one year of entry. Patients on methadone programs are not excluded.

4.3.16 Inability to abstain from alcohol throughout the entire course of treatment and follow-up.

4.3.17 History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease.

4.3.18 History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
evaluate the safety, tolerability, and efficacy of Peginterferon a-2a plus Ribavirin for the treatment of chronic hepatitis C (CHC) infection in persons co-infected with human immunodeficiency virus (HIV) who have failed to achieve a sustained virologi

SECONDARY OUTCOMES:
To evaluate the virological response at weeks 12 and 24 as compared to baseline values.
To evaluate the sustained virological response at post-treatment weeks 4, 12, and 24 as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dieterich, MD, Principal Investigator — Chair - Hepatitis Resource Network
Locations (1):
- Mt. Sinai School of Medicine, New York, New York, United States